CLINICAL TRIAL: NCT06555380
Title: Impact of Multifactorial Lifestyle Interventions on Psychosocial Well-being for Children Living With Obesity
Brief Title: Childhood Obesity, Lifestyle Interventions and Psychosocial Well-being
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus Municipality, Denmark (Other); Randers Municipality, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: 3518
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Pediatric Obesity; Psychosocial Well-being
Keywords: Lifestyle Intervention; Pediatric Obesity; Psychosocial Well-being; Long-term impact
MeSH Terms: conditions — Pediatric Obesity | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- The one-year intervention group: Children aged 5-10 with obesity who participated in the one-year multifactorial family-centered lifestyle intervention.
  Interventions: Behavioral: The one-year intervention
- The three-year intervention group: Children aged 5-10 with obesity who participated in the three-year multifactorial family-centered lifestyle intervention.
  Interventions: Behavioral: The three-year intervention
- The non-intervention group: Children with obesity living in one of the municipalities who were never invited to participate in the interventions.

INTERVENTIONS:
Behavioral: The one-year intervention — A multifactorial family-centered lifestyle intervention with a maximum duration of one year, corresponding to three-four visits. Participants were offered complimentary weekly supervised physical activity. The day-to-day intervention was managed by specialized nurses at local healthcare centers, at the participants' homes, or in a local clinic.
  Groups: The one-year intervention group
Behavioral: The three-year intervention — A multifactorial family-centered lifestyle intervention extending up to three years, with clinical visits at local healthcare centers which included repeatedly visits (up to 8 times / year). The intervention was managed by specialized nurses.
  Groups: The three-year intervention group

SUMMARY:
Childhood obesity has been associated with an increased risk of impaired psychosocial well-being and the development of depression and anxiety.

This study includes approximately 200 children with obesity aged 5-10 treated within one of two multifactorial family-centered lifestyle intervention in the time-period 2014-2020. Additionally, this study includes 150 children with obesity in the same age group, who were never invited into the multifactorial family-centered lifestyle interventions. During that period the children annually completed the Danish Nation Well-being Questionnaire (DNWQ) in school. The DNWQ is a national questionnaire used to examine the well-being and learning environment in Danish schoolchildren.

The aim is to investigate the long-term impact on psychosocial well-being in children with obesity following participation in one of two multifactorial family-centered lifestyle interventions: a one-year and three-year intervention. Further, to compare this alteration in psychosocial well-being between the intervention groups and with a reference group of children who were never invited to participate in the interventions.

The study will combine data from mandatory health check-ups at school, the Danish National Registries, and the Danish agency for IT and Learning (STIL), The ministry of Education.

DETAILED DESCRIPTION:
The continuous rise in obesity among children has become a critical public health issue, due to the associated risks of continuous obesity and development of metabolic disorders in adulthood. While these consequences may not become apparent until later in life, the obesity-related complications commonly observed in childhood are associated with impaired psychosocial well-being (i.e. reduced self-image, bullying, and stigmatization). Children and adolescents with obesity have a higher risk of impaired health-related quality of life (QoL) and are more likely to suffer from depression and anxiety, compared to their lean peers. Furthermore, these mental health related complications can typical be observed in childhood opposite the somatic complications.

While there is agreement that obesity is associated with overall reduced psychosocial well-being in children and adolescents, studies comparing how different, or no lifestyle interventions affects psychosocial well-being remain scarce. It is therefore necessary to identify effective lifestyle interventions, that can handle and improve this issue.

The aim of this study is therefore to investigate the long-term impact on psychosocial well-being in children with obesity following participation in one of two multifactorial family-centered lifestyle interventions: a one-year and a three-year intervention. Further, to compare this alteration in psychosocial well-being between the intervention groups and with a reference group of children who were never invited to participate in the interventions. Additionally, the study aims to eliminate the potential impact of weight change on the association between exposure and change in psychosocial well-being.

Study design: This observational cohort study will combine data from obligatory health check-ups at school, the Danish National Registries, and the Ministry of Education for children aged 5-10 with obesity living in two municipalities in Denmark between August 1st, 2014, and June 30th, 2020. The last possible day of follow-up will be February 1st, 2023.

The interventions:

The one-year intervention: A multifactorial family-centered lifestyle intervention offering a maximum duration of one year, corresponding to three-four visits. Participants were offered complimentary weekly supervised physical activity. The day-to-day intervention was managed by specialized health care nurses at local treatment centers, at the participants' homes, or in a local clinic.

The three-year intervention: A multifactorial family-centered lifestyle intervention extending up to three years, with clinical visits at local healthcare centers occurring approximately every eight weeks, managed by specialized nurses.

The participants:

Children in the intervention groups were 5 to 10 years of age and participated in one of two different family-centered interventions: a one-year or three-year intervention. Children with obesity living in one of the municipalities, who were never invited to participate in the interventions will act as a reference group for this study. The inclusion visit for this group is defined as the initial observation with obesity.

Obesity will be defined by the International Obesity Task Force (IOTF) guideline as a BMI >= 30 kg/m2 adjusted for age and sex.

The following children will be included in this trial:

* 107 children with obesity treated with the one-year intervention
* 66 children with obesity treated with the three-year intervention
* 146 children with obesity who were not invited to participate in the interventions (non intervention group)

Data-collection and analyses:

Children who participated in one of the two interventions will be identified by using data from TM-Sund and NOVAX. Data recorded at health check-ups at the school containing height and weight will also be extracted from TM-Sund and NOVAX. TM-Sund and NOVAX are data capturing tools used by the community health care nurses employed at the two municipalities. The reference group will be identified in TM-Sund.

The DNWQ data will be obtained from the Danish agency for IT and Learning (STIL), The ministry of Education.

Data on socioeconomic status (SES), immigration, family structure, and psychiatric diagnoses will be obtained from the national Danish registries through Statistics Denmark.

Ethics & Permissions:

The local committee on health ethics have approved the overall project and data transfer (rec.no 1-45-70-27-20). The project is internally reported to the University of Aarhus (rec no. 3518). The project has achieved approval from The Danish Data Protection Agency and the Principal Investigator has been granted accessed to data from registers from Danish Statistics.

The researchers have no conflict of interest to declare.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion visit between August 1st, 2014, and June 30th, 2020.
* Obesity at time of referral as defined by the IOTF guideline as a BMI >= 30 kg/m2 adjusted for age and sex.
* Obesity at time of referral as defined by the IOTF guideline as a BMI >= 30 kg/m2 adjusted for age and sex.
* Age between 5 and 10 years at inclusion visit.
* A completed DNWQ within a timeframe of 10 months prior to 2 months after inclusion.
* A completed DNWQ at follow-up (1 to 3 years after inclusion visit).

Exclusion Criteria:

* Children declining participation in a community-based lifestyle intervention.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with obesity, 5-10 years of age living in two municipalities in Denmark between August 1st, 2014, and June 30th, 2020. The children have either received treatment with one of the multifactorial family-centered lifestyle interventions or where never invited into the interventions.
Sampling Method: Non-Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change in psychosocial well-being as assessed by the DNWQ, obtained from the Danish agency for IT and Learning (STIL), The ministry of Education. | Annually from August 1st, 2014, to February 1st, 2023)
  The impact on psychosocial well-being will be assessed with responses to specific questions regarding psychosocial well-being related to school from the DNWQ at time of inclusion and at follow-up.
  The DNWQ is a national questionnaire completed annually in primary school and used to examine how primary schoolchildren perceive their well-being and learning environment in school.
  The following four questions have been selected as our primary outcomes.
  1. Question:
     Are you happy with your school?
  2. Questions:
     Do you feel lonely at school? (0-3 grade) Do you feel lonely? (4-9 grade)
  3. Question:
     Is anyone teasing you so that you feel sad? (0-3 grade) Have you been bullied this school year? (4-9 grade)
  4. Question:
  Does your stomach ache when you are at school? (0-3 grade) How often does your stomach ache? (4-9 grade)

SECONDARY OUTCOMES:
Change in psychosocial well-being as assessed by the DNWQ, obtained from the Danish agency for IT and Learning (STIL), The ministry of Education. | Annually from August 1st, 2014, to February 1st, 2023)
  Same as primary outcome measure, but with other questions chosen from the DNWQ.
  The following three questions has been selected as our secondary outcome.
  A. Question:
  Are you good at solving your problems? (0-3 grade) How often can you find a solution to problems, just by trying hard enough? (4-9 grade)
  B. Question:
  Can you concentrate during class?
  C. Question:
  Are you good at helping each other in class? (0-3 grade) Most students in my class are friendly and helpful. (4-9 grade)

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Participant data (IPD) will be available on reasonable request.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT06555380/Prot_SAP_000.pdf